CLINICAL TRIAL: NCT01198626
Title: A Randomized, Controlled, Double Blind, Multicenter, Phase 2 Study of the Safety/Tolerability and Efficacy of JNJ-32729463 Compared With Moxifloxacin for the Treatment of Subjects Requiring Hospitalization for Community-Acquired Bacterial Pneumonia (CABP) With a PORT Score of II or Greater
Brief Title: Efficacy and Safety Study of JNJ-32729463 Compared With Moxifloxacin for the Treatment of Subjects Requiring Hospitalization for Community-Acquired Bacterial Pneumonia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment would not have been met prior to the end of the pneumonia season. Termination is based on slow enrollment and not related to safety or efficacy.
Sponsor: Furiex Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 32729463CAP2001
Record Dates: First submitted 2010-09-07; First posted 2010-09-10 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Community-Acquired Bacterial Pneumonia (CABP)
Keywords: community-acquired bacterial pneumonia; CABP; CAP; pneumonia; pneumonia, bacterial; bacterial infections; anti-bacterial agents; anti-infective agents; lung disease, interstitial; respiratory tract diseases; respiratory tract infections; community-acquired infections
MeSH Terms: conditions — Pneumonia; Pneumonia, Bacterial; Bacterial Infections; Lung Diseases, Interstitial; Respiratory Tract Diseases; Respiratory Tract Infections; Community-Acquired Infections | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- JNJ-32729463 (Experimental)
  Interventions: Drug: JNJ-32729463
- moxifloxacin (Active Comparator)
  Interventions: Drug: moxifloxacin
- JNJ-32729463 Open-Label (Experimental): subjects with suspected or confirmed S. aureus CABP may be entered into an open-label JNJ 32729463 treatment group at selected study sites
  Interventions: Drug: JNJ-32729463 (Open-Label)

INTERVENTIONS:
Drug: JNJ-32729463 — 150 mg intravenous formulation administered twice daily for at least 72 hours, followed by 250 mg oral formulation administered twice daily for a total treatment time of 7 to 14 days
  Arms: JNJ-32729463
Drug: moxifloxacin — 400 mg intravenous formulation administered once daily for at least 72 hours, followed by 400 mg oral formulation administered once daily for a total treatment time of 7 to 14 days. To maintain the blind, subjects will receive one dose of moxifloxacin and one dose of placebo daily.
  Other Names: Avelox
  Arms: moxifloxacin
Drug: JNJ-32729463 (Open-Label) — Subjects may receive JNJ-32729463 intravenous formulation up to 150 mg either BID or TID followed by 250 mg oral formulation BID for a total treatment time of 7 to 14 days.
  Arms: JNJ-32729463 Open-Label

SUMMARY:
The purpose of this study is to determine the efficacy, safety and tolerability of JNJ-32729463 compared to moxifloxacin for the treatment of subjects requiring hospitalization for Community-Acquired Bacterial Pneumonia (CABP).

ELIGIBILITY:
Inclusion Criteria:

* women of childbearing potential must agree to use an acceptable method of birth control
* clinical diagnosis of community acquired bacterial pneumonia (CABP)
* PORT score of II or greater
* able to generate an adequate sputum specimen
* chest x-ray showing presence of new infiltrates in a lobar or multilobar distribution characteristic of bacterial pneumonia

Exclusion Criteria:

* history of tendon damage/disorders due to quinolone therapy
* uncorrected hypokalemia
* history of myasthenia gravis
* intubated at the time of consent OR subject is a candidate for enrollment into the open-label S. aureus arm and has been intubated greater than 12 hours prior to randomization
* mild CABP with a PORT score of less than II
* viral, fungal, mycobacterial, or atypical pneumonia as a primary diagnosis
* pneumonia suspected to be secondary to aspiration
* primary, solitary lung abscess
* healthcare-associated pneumonia, hospital-acquired pneumonia, or ventilator-associated pneumonia
* known bronchial obstruction or a history of postobstructive pneumonia.
* primary lung cancer or another malignancy metastatic to the lungs
* cystic fibrosis, known or suspected Pneumocystis jiroveci (carinii) pneumonia, or known or suspected active tuberculosis
* infection that necessitates the use of a concomitant antibacterial agent in addition to study medication
* systemic antibiotics within the last 96 hours before randomization, with exceptions
* hospitalized for greater than 72 hours for any reason 30 days before randomization (excluding the 24 hour period before enrollment).
* history of a serious hypersensitivity reaction to any quinolone including moxifloxacin.
* female and pregnant, breastfeeding, or may be pregnant.

Other protocol-specific eligibility criteria may apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Resolution of signs and symptoms of community-acquired bacterial pneumonia | Day 19 (Test of Cure Visit)

SECONDARY OUTCOMES:
Daily signs and symptoms of CABP | Up to Day 19
Microbiological response: per-pathogen and per-subject | Day 19 (Test of Cure Visit)
Percent of subjects with resolution of signs and symptoms of CABP | Day 3 and Day 4
Clinical outcome in subjects with S. pneumoniae | Day 19 (Test of Cure Visit)
Rate of superinfections or new infections | Day 30
Time to oral switch | Day 14
All-cause mortality | Up to Day 30

CONTACTS AND LOCATIONS:
Locations (32):
- United States (11):
  - Furiex Research Site, Mobile, Alabama
  - Furiex Research Site, Sylmar, California
  - Furiex Research Site, Orlando, Florida
  - Furiex Research Site, Vero Beach, Florida
  - Furiex Research Site, Peoria, Illinois
  - Furiex Research Site, Hazard, Kentucky
  - Furiex Research Site, Anaconda, Montana
  - Furiex Research Site, Omaha, Nebraska
  - Furiex Research Site, Albueuerque, New Mexico
  - Furiex Research Site, Austin, Texas
  - Furiex Research Site, Longview, Washington
- Canada (3):
  - Furiex Research Site, Calgary, Alberta
  - Furiex Research Site, Chicoutimi, Quebec
  - Furiex Research Site, Québec, Quebec
- Colombia (2):
  - Furiex Research Site, Bogotá
  - Furiex Research Site, Cali
- Germany (5):
  - Furiex Research Site, Greifswald
  - Furiex Research Site, Hanover
  - Furiex Research Site, Hofheim
  - Furiex Research Site, Homburg/Saar
  - Furiex Research Site, Paderborn
- Hungary (5):
  - Furiex Research Site, Csorna
  - Furiex Research Site, Debrecen
  - Furiex Research Site, Gyöngyös
  - Furiex Research Site, Miskolc
  - Furiex Research Site, Tatabánya
- Poland (6):
  - Furiex Research Site, Bialystok
  - Furiex Research Site, Bydgoszcz
  - Furiex Research Site, Bystra
  - Furiex Research Site, Lodz
  - Furiex Research Site, Skierniewice
  - Furiex Research Site, Warsaw